CLINICAL TRIAL: NCT05143619
Title: Impact of "Teaching the Teachers" Concept on Global Education and Application of Hepatocellular Carcinoma Diagnosis Guidelines
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2018-1157; NCI-2021-10961 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-1157 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-11-18; First posted 2021-12-03 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (surveys): Participants complete surveys immediately after completion of a HCC diagnostic guideline webinar, monthly thereafter, and again at 6 months.
  Interventions: Other: Survey Administration

INTERVENTIONS:
Other: Survey Administration — Complete surveys

SUMMARY:
This study evaluates a concept called 'Teaching the Teachers' and whether it is helpful in disseminating guidelines on the national and international levels. "Teaching the Teachers" involves teaching the guidelines to experts who later teach the same guidelines to other radiologists, trainees, and physicians to assume the teacher's role and disseminate the guidelines and so on.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the magnitude of teaching of hepatocellular carcinoma (HCC) diagnostic guidelines after applying "Teaching the Teachers" concept.

II. Assess the effect of "Teaching the Teachers" concept on application of guidelines in clinical practice.

OUTLINE:

Participants complete surveys immediately after completion of a HCC diagnostic guideline webinar, monthly thereafter, and again at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Physicians who finished radiology residency
* Radiologists with current or completed specialized training in abdominal imaging
* Radiologists with expertise in liver imaging with no minimum number of years of experience
* Radiologists working in academic, community, and governmental practices
* Radiologists with current practice in any country around the globe
* Radiologists with and without previous knowledge of HCC diagnosis guidelines (Liver Imaging Reporting and Data System [LI-RADS])
* Radiologists with interest in education and/or teaching

Exclusion Criteria:

* Physicians with no formal training in radiology
* Radiologists with no expertise in abdominal/liver imaging
* Current radiology residents
* Radiologists with no interest in education and/or teaching

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Abdominal radiologists with expertise in liver imaging working in academic, community, and governmental practices in many centers around the world.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-05-10 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Teaching rates of the hepatocellular carcinoma diagnosis guidelines | Through study completion, an average of 1 year
  Paired comparisons will be performed on the proportion of learners using the practice guidelines. Will perform a multivariate analysis to assess the effect of demographic characteristics (e.g., number of years of experience, type of practice) on the teaching rate of the HCC diagnostic guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Khaled M Elsayes, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Anderson Cancer Center — http://www.mdanderson.org